CLINICAL TRIAL: NCT00208910
Title: A Study of Enhancement of Progressive Muscle Relaxation Therapy for Generalized Anxiety Disorder Through Use Of An Odorant Cue.
Brief Title: Muscle Relaxation Therapy With Odorant Cue
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 0860-2003
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2013-11-11 (Estimated); Status verified 2013-11

CONDITIONS: Generalized Anxiety Disorder; Anxiety
Keywords: Anxiety; Mental Health
MeSH Terms: conditions — Generalized Anxiety Disorder; Anxiety Disorders; Psychological Well-Being

INTERVENTIONS:
Behavioral: Odorant Cue

SUMMARY:
A novel procedure for generalized anxiety disorder where an odorant cue is paired with the state of deep relaxation during training. It is hypothesized that by smelling the odor in an anxiety-provoking situation, the patient will more easily invoke a state of relaxation, providing greater relief from the distressing tension and worry that characterize GAD.

DETAILED DESCRIPTION:
We hypothesize that by presenting a novel odor to a patient in a state of deep relaxation, the odor will serve as a conditioned inhibitory stimulus, or safety signal, in anxiety-provoking situations. With the odor serving as a contextual cue for the state of relaxation.

ELIGIBILITY:
Inclusion Criteria:

* GAD without a comorbid active major psychiatric disorder.
* GAD must be the primary active psychiatric disorder.
* GAD determined via the Mini International Neuropsychiatric Interview (MINI).

Exclusion Criteria:

* Significant medical illness that might interfere with the relaxation therapy or with training using the odorant.
* Actively abusing alcohol.
* Illicit substances.
* Currently using rapid-acting anxiolytic agents (e.g. benzodiazepines, hydroxyzine).
* Started an antidepressant, antipsychotic or mood stabilizing agent within three months of screening visit.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15
Dates: Start 2003-11; Study Completion 2005-05

PRIMARY OUTCOMES:
PSWQ

SECONDARY OUTCOMES:
HAM-A

CONTACTS AND LOCATIONS:
Overall Officials: Philip T Ninan, MD, Principal Investigator — Emory University
Locations (1):
- Emory University School of Medicine, Atlanta, Georgia, United States